CLINICAL TRIAL: NCT04476914
Title: Psychological Distress Symptoms in Family Members of Patients With COVID-19 Respiratory Failure in Intensive Care Units
Brief Title: Stress Related Disorders in Family Members of COVID-19 Patients Admitted to the ICU
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Washington (Other); Tulane University (Other); University of Vermont (Other); Penn State University (Other); Columbia University (Other); South Shore Hospital (Other); Evergreen Hospital (Unknown); Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20-1021
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Failure; SARS-CoV 2; Corona Virus Infection; Post Intensive Care Unit Syndrome; Family Members; Post Traumatic Stress Disorder; Anxiety; Depression
MeSH Terms: conditions — Respiratory Insufficiency; Coronavirus Infections; Stress Disorders, Post-Traumatic; Anxiety Disorders; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Family Member: Family members of ICU patients admitted with respiratory failure from COVID-19

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a novel infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). This syndrome has been associated with high mortality, estimated to be about 1.7% of all infected in the US, though in those who develop acute respiratory distress syndrome (ARDS) in the context of the infection, mortality rates appear to be much higher, perhaps up to 70%. To avoid transmission of the virus, patient isolation has become the standard of care, with many hospitals eliminating visitors of any type, and particularly eliminating visitation to patients infected with COVID-19. These necessary, but restrictive, measures add stress to the ICU and particularly to the family members who are not only left with fear, but also many unanswered questions. In contrast to the Society of Critical Care Guidelines (SCCM) which recommend family engagement in the ICU and recent data from this study team which suggests engaging families in end-of-life situations reduces symptoms of Post-Traumatic Stress Disorder (PTSD) in family members, family members are now unable to say good-bye and unable to provide support to their loved-one throughout the process of the patients' ICU stay. The study hypothesizes is that these restrictive visiting regulations will increase rates of Post-intensive care syndrome- family (PICS-F) which includes symptoms of PTSD, depression, and anxiety and aim to evaluate for factors that either exacerbate these symptoms or protect from them.

DETAILED DESCRIPTION:
The study aims to define the prevalence of PICS-F in the study population 3-4 months after ICU admission of patient, specifically symptoms of PTSD as the primary outcome, and symptoms of depression and anxiety as secondary outcomes. The study hypothesizes prevalence will be higher than seen in other studies.

An additional aim is to identify predisposing or mitigating exposures for PICS-F. The study hypothesizes that increased psychological symptoms will be associated less exposure to virtual patient visits (tablet/video conferencing), higher number of patient comorbidities (using the Charleston comorbidity index), preexisting family member psychological conditions.

The study also plans to evaluate the association between family perception of quality of communication or decision-making using items from the validated Family Satisfaction in the ICU (FS-ICU) and psychological symptoms. The study hypothesizes that the quality of communication and decision-making will be associated with lower psychological symptoms.

Finally, the plan is to, using qualitative methods, explore and describe family members' stress, experiences with communication with healthcare providers and their satisfaction with ICU care while being physically distant from their loved ones. The aim is to use qualitative findings about family members' experiences to contextualize and explain results differences in stress, satisfaction and communication quality between low vs high PICS-F scores.

ELIGIBILITY:
Inclusion Criteria:

* Family members of COVID-19 positive patients admitted to the Intensive Care Unit with respiratory failure

Exclusion Criteria:

* Family members will be excluded if they: are under 18 or unable to complete the survey's due to language barriers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be consenting family members of COVID-19 positive patients who are admitted to the intensive care unit with respiratory failure
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Symptoms of Post-Traumatic Stress Disorder (PTSD) | 90-120 days after admission of patient to the ICU
  Using Impact of Events Scale-Revised-6 , family members will be screened for symptoms of PTSD. Scale returns scores of 0-24, with higher scores indicating more likely to have symptoms of PTSD

SECONDARY OUTCOMES:
Symptoms of Anxiety | 90-120 days after admission of patient to the ICU
  Using the Hospital Anxiety and Depression Score, family members will be screened for symptoms of anxiety. The HADS anxiety scale is scored between 0 and 21, with higher scores indicating more likely to have symptoms of anxiety
Symptoms of Depression | 90-120 days after admission of patient to the ICU
  Using the Hospital Anxiety and Depression Score, family members will be screened for symptoms of Depression. The HADS depression scale is scored between 0 and 21, with higher scores indicating more likely to have symptoms of depression
Family Satisfaction with Communication and Decision Making | 90-120 days after admission of patient to the ICU
  Using preselected questions from the Family Satisfaction in the ICU-27 questionnaire, we will survey families to evaluate their satisfaction with communication and decision making. Higher scores will indicate more satisfication

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Eastern Colorado Veterans Affairs Health Care System, University Of Colorado, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Tulane Medical Center, New Orleans, Louisiana
  - Brigham and Women's Medical Center, Boston, Massachusetts
  - South Shore Medical Center, Weymouth, Massachusetts
  - Columbia Milstein and Allen Hospitals, New York, New York
  - Penn State Hershey Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] https://www.cdc.gov/coronavirus/2019-ncov/cases-updates/cases-in-us.html. Accessed on 3/30/2020
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Davidson JE, Aslakson RA, Long AC, Puntillo KA, Kross EK, Hart J, Cox CE, Wunsch H, Wickline MA, Nunnally ME, Netzer G, Kentish-Barnes N, Sprung CL, Hartog CS, Coombs M, Gerritsen RT, Hopkins RO, Franck LS, Skrobik Y, Kon AA, Scruth EA, Harvey MA, Lewis-Newby M, White DB, Swoboda SM, Cooke CR, Levy MM, Azoulay E, Curtis JR. Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU. Crit Care Med. 2017 Jan;45(1):103-128. doi: 10.1097/CCM.0000000000002169. PMID 27984278
- [Background] Amass TH, Villa G, OMahony S, Badger JM, McFadden R, Walsh T, Caine T, McGuirl D, Palmisciano A, Yeow ME, De Gaudio R, Curtis JR, Levy MM. Family Care Rituals in the ICU to Reduce Symptoms of Post-Traumatic Stress Disorder in Family Members-A Multicenter, Multinational, Before-and-After Intervention Trial. Crit Care Med. 2020 Feb;48(2):176-184. doi: 10.1097/CCM.0000000000004113. PMID 31939785
- [Background] Davidson JE, Jones C, Bienvenu OJ. Family response to critical illness: postintensive care syndrome-family. Crit Care Med. 2012 Feb;40(2):618-24. doi: 10.1097/CCM.0b013e318236ebf9. PMID 22080636
- [Background] Lautrette A, Darmon M, Megarbane B, Joly LM, Chevret S, Adrie C, Barnoud D, Bleichner G, Bruel C, Choukroun G, Curtis JR, Fieux F, Galliot R, Garrouste-Orgeas M, Georges H, Goldgran-Toledano D, Jourdain M, Loubert G, Reignier J, Saidi F, Souweine B, Vincent F, Barnes NK, Pochard F, Schlemmer B, Azoulay E. A communication strategy and brochure for relatives of patients dying in the ICU. N Engl J Med. 2007 Feb 1;356(5):469-78. doi: 10.1056/NEJMoa063446. PMID 17267907
- [Background] Azoulay E, Pochard F, Kentish-Barnes N, Chevret S, Aboab J, Adrie C, Annane D, Bleichner G, Bollaert PE, Darmon M, Fassier T, Galliot R, Garrouste-Orgeas M, Goulenok C, Goldgran-Toledano D, Hayon J, Jourdain M, Kaidomar M, Laplace C, Larche J, Liotier J, Papazian L, Poisson C, Reignier J, Saidi F, Schlemmer B; FAMIREA Study Group. Risk of post-traumatic stress symptoms in family members of intensive care unit patients. Am J Respir Crit Care Med. 2005 May 1;171(9):987-94. doi: 10.1164/rccm.200409-1295OC. Epub 2005 Jan 21. PMID 15665319
- [Background] Wall RJ, Engelberg RA, Downey L, Heyland DK, Curtis JR. Refinement, scoring, and validation of the Family Satisfaction in the Intensive Care Unit (FS-ICU) survey. Crit Care Med. 2007 Jan;35(1):271-9. doi: 10.1097/01.CCM.0000251122.15053.50. PMID 17133189
- [Background] Sundin EC, Horowitz MJ. Horowitz's Impact of Event Scale evaluation of 20 years of use. Psychosom Med. 2003 Sep-Oct;65(5):870-6. doi: 10.1097/01.psy.0000084835.46074.f0. PMID 14508034
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Curtis JR, Treece PD, Nielsen EL, Gold J, Ciechanowski PS, Shannon SE, Khandelwal N, Young JP, Engelberg RA. Randomized Trial of Communication Facilitators to Reduce Family Distress and Intensity of End-of-Life Care. Am J Respir Crit Care Med. 2016 Jan 15;193(2):154-62. doi: 10.1164/rccm.201505-0900OC. PMID 26378963
- [Background] Carson SS, Cox CE, Wallenstein S, Hanson LC, Danis M, Tulsky JA, Chai E, Nelson JE. Effect of Palliative Care-Led Meetings for Families of Patients With Chronic Critical Illness: A Randomized Clinical Trial. JAMA. 2016 Jul 5;316(1):51-62. doi: 10.1001/jama.2016.8474. Erratum In: JAMA. 2017 May 23;317(20):2134. doi: 10.1001/jama.2017.4298. PMID 27380343
- [Background] White DB, Angus DC, Shields AM, Buddadhumaruk P, Pidro C, Paner C, Chaitin E, Chang CH, Pike F, Weissfeld L, Kahn JM, Darby JM, Kowinsky A, Martin S, Arnold RM; PARTNER Investigators. A Randomized Trial of a Family-Support Intervention in Intensive Care Units. N Engl J Med. 2018 Jun 21;378(25):2365-2375. doi: 10.1056/NEJMoa1802637. Epub 2018 May 23. PMID 29791247
- [Background] Van Scoy LJ, Chiarolanzio PJ, Kim C, Heyland DK. Development and initial evaluation of an online decision support tool for families of patients with critical illness: A multicenter pilot study. J Crit Care. 2017 Jun;39:18-24. doi: 10.1016/j.jcrc.2016.12.022. Epub 2017 Jan 19. No abstract available. PMID 28131020
- [Background] Heyland DK, Davidson J, Skrobik Y, des Ordons AR, Van Scoy LJ, Day AG, Vandall-Walker V, Marshall AP. Improving partnerships with family members of ICU patients: study protocol for a randomized controlled trial. Trials. 2018 Jan 4;19(1):3. doi: 10.1186/s13063-017-2379-4. PMID 29301555